CLINICAL TRIAL: NCT04648969
Title: Prolonged Pulsatile Kisspeptin Administration in Hypogonadotropic Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stephanie B. Seminara, MD (Other)
Responsible Party: Sponsor-Investigator, Stephanie B. Seminara, MD, Chief, Reproductive Endocrine Unit; Massachusetts General Hospital; Professor of Medicine, Harvard Medical School; Director, MGH Harvard Center for Reproductive Medicine, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 313509
Record Dates: First submitted 2020-11-11; First posted 2020-12-02 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hypogonadotropic Hypogonadism
Keywords: hypogonadotropic hypogonadism, kisspeptin
MeSH Terms: conditions — Hypogonadism | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: kisspeptin, GnRH (Experimental): • Intravenous administration of kisspeptin 112-121; 20 boluses in a 40-hour period. Intravenous administration of GnRH; one bolus.
  Interventions: Drug: kisspeptin 112-121; Drug: GnRH

INTERVENTIONS:
Drug: kisspeptin 112-121 — 20 intravenous doses of kisspeptin 112-121 (4 different doses of kisspeptin (randomized) in 5 sets)
  Other Names: metastin 45-54
Drug: GnRH — 1 intravenous dose of GnRH
  Other Names: gonadotropin-releasing hormone

SUMMARY:
The goal of this study is to develop novel treatments for patients with a condition called hypogonadotropic hypogonadism (HH) through the use of exogenous kisspeptin.

DETAILED DESCRIPTION:
* Assignment: Each study subject will serve as their own control. The order of kisspeptin doses will be randomized within each set/exposure.
* Delivery of Interventions:

  * Prior to the study visit, subjects will undergo a review of their medical history and screening laboratories. Subjects will also wear a gonadotropin releasing hormone (GnRH) pump prior to the inpatient study visit.
  * On the day of the inpatient study, the subjects will

    * Undergo q10 min blood sampling for 6 hours,
    * Receive kisspeptin intravenous (IV) boluses from hour 6 to hour 44 (20 boluses total),
    * Undergo q10 min blood samplings for another 6 hours,
    * Receive a single GnRH IV bolus at hour 51.

ELIGIBILITY:
Inclusion/exclusion criteria:

* Age 18 years and older,
* Confirmed diagnosis of HH with

  * Low testosterone or estradiol,
  * Low or low-normal gonadotropin levels,
  * Thyroid stimulating hormone (TSH) and prolactin within the reference range,
  * Absence of abnormal pituitary or hypothalamic findings on Magnetic resonance imaging (MRI),
* All other medical conditions stable and well controlled,
* No prescription medications known to affect reproductive endocrine function for at least 2 months or for 5 half-lives of the drug (whichever is shorter) except for medications used to treat the subject's reproductive condition,
* No history of a medication reaction requiring emergency medical care,
* No illicit drug use,
* No excessive alcohol consumption (<10 drinks/week),
* Normal blood pressure (BP), (systolic BP < 140 mm Hg, diastolic < 90 mm Hg),
* White blood cell, platelet counts, and TSH between 90% of the lower limit and 110% of the upper limit of the reference range,
* Prolactin below 110% of the upper limit of the reference range,
* Hemoglobin

  * Women: no less than 0.5 gm/dL below the lower limit of the reference range for normal women,
  * Men: on adequate testosterone replacement therapy: normal male reference range,
* Blood urea nitrogen (BUN), creatinine, aspartate aminotransferase (AST), alanine transaminase (ALT) not elevated,
* For women,

  * Negative serum human chorionic gonadotropin (hCG) pregnancy test at the time of screening (additional urine pregnancy test will be conducted prior to drug administration),
  * Not breastfeeding and not pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Average change in luteinizing hormone (LH) pulse amplitude in response to kisspeptin | 52 hours
  Change in LH amplitude before, during and after kisspeptin administration

SECONDARY OUTCOMES:
Average change in LH pulse frequency in response to kisspeptin | 52 hours
  Change in LH frequency before and after kisspeptin administration

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Seminara, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No